CLINICAL TRIAL: NCT02070250
Title: Examination of a Stress Management Intervention for Cancer Patients as Delivered by Community Mental Health Professionals
Brief Title: Stress Management for Cancer Patients: How Well Does it Work? (C2H-D)
Acronym: C2H-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Andersen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-13127; R25CA163197 (NIH)
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Mood; Stress, Psychological
Keywords: Stress management; Coping skills; Recently diagnosed cancer patients; Intervention, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- From Cancer to Health (C2H-D) (Experimental): Individuals participating in the From Cancer to Health (C2H-D) Stress Management Psychological Intervention
  Interventions: Behavioral: From Cancer to Health (C2H-D)

INTERVENTIONS:
Behavioral: From Cancer to Health (C2H-D) — From Cancer to Health gives people with cancer the information and tools they need to manage their stress to improve their health throughout the cancer journey. Each institution involved in this study will implement the core techniques of the C2H-D Intervention but may alter the format somewhat to meet their patient population needs (e.g., shorten hourly 18 week intervention into 2-hour 9 week intervention).
  Other Names: C2H; Biobehavioral Intervention; BBI; Stress management

SUMMARY:
Psychological interventions for cancer patients have been tested and found to reduce stress and improve quality of life. These interventions have been tested at academic medical centers but have not been available for use by community mental health professionals. One such intervention is the Biobehavioral Intervention (BBI), developed by Professor Barbara L. Andersen and colleagues at Ohio State (OSU). Current funding has enabled the investigators to train mental health professionals from across the country to deliver the BBI at their institution. Recently diagnosed cancer patients who are participating in the BBI group at these institutions may participate in a research study completing self report measures asking about psychological and behavioral outcomes (for example, mood, stress, diet and physical activity). The investigators hypothesize that individuals participating in the intervention will report improvements in outcomes, such as reduced stress and improved mood, reduced symptoms of the disease and treatment, etc., after completing the intervention and continue to report these improvements up to 6 months after the group ends. OSU will coordinate this data collection project but information about participating sites is listed in http://clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Recent initial diagnosis of cancer without metastatic disease
* Able to speak/read English

Exclusion Criteria: Those with concurrent diagnoses of

* Organic brain syndrome
* Dementia
* Mental retardation
* non-English speaking
* Significant sensory deficit
* Severe mental illness (e.g., schizophrenia, psychotic disorder)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-11; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post-intensive intervention assessment in mood on the 65-item Profile of Mood States (POMS) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.
Change from baseline to post-intensive intervention assessment in cancer-specific stress on the 20-item Impact of Events Scale (IES) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.

SECONDARY OUTCOMES:
Change from baseline to post-intensive intervention assessment in social support using the 20 item Perceived Social Support from Your Family Scale (PSS-Fa) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.
Change from baseline to post-intensive intervention assessment in physical activity on the 3-item Physical Activity Rating Scale (PAR) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.
Change from baseline to post-intensive intervention assessment in diet on the 23-item Food Habits Questionnaire (FHQ) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.
Change from baseline to post-intensive intervention assessment in sexual health on the 4-item Your Sexual Life questionnaire | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.

OTHER OUTCOMES:
Change from baseline to post-intensive intervention assessment in pain using the 13-item Brief Pain Questionnaire (BPQ) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.
Change from baseline to post-intensive intervention assessment in fatigue using the 7-item Fatigue Severity Index (FSI) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.
Change from baseline to post-intensive intervention assessment in sleep using the 24-item Pittsburgh Sleep Quality Index (PSQI) | Baseline, up to 18 weeks
  The intensive intervention length can vary by location from 4 to 18 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Andersen, PhD, Principal Investigator — Ohio State University
Locations (15):
- United States (15):
  - Cancer Center of East Alabama Medical Center, Auburn, Alabama
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Wellness House, Hinsdale, Illinois
  - Cancer Wellness Center, Northbrook, Illinois
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Genesis Health Center, Davenport, Iowa
  - Unity Point Health/Gilda's Club Quad Cities, Davenport, Iowa
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - OSU Stephanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Seton UT Southwestern, Austin, Texas
  - Baylor Regional Medical Center at Plano, Texas, Plano, Texas

REFERENCES:
- [Background] Ashmore JA, Ditterich KW, Conley CC, Wright MR, Howland PS, Huggins KL, Cooreman J, Andrews PS, Nicholas DR, Roberts L, Hewitt L, Scales JN, Delap JK, Gray CA, Tyler LA, Collins C, Whiting CM, Brothers BM, Ryba MM, Andersen BL. Evaluating the effectiveness and implementation of evidence-based treatment: A multisite hybrid design. Am Psychol. 2019 May-Jun;74(4):459-473. doi: 10.1037/amp0000309. Epub 2018 Jul 19. PMID 30024215